CLINICAL TRIAL: NCT00924781
Title: A Phase II Randomized, Open-Label, Multiple-Rising Dose Clinical Trial to Study the Efficacy and Safety of MK2578 for the Maintenance of Anemia Treatment in Patients With Chronic Kidney Disease Who Are on Hemodialysis.
Brief Title: A Study of the Efficacy and Safety of MK2578 for the Treatment of Anemia in Patients With Kidney Disease (MK2578-003-AM03-EXT12)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2578-003; 2009_603
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Anemia associated with chronic kidney disease (CKD); Hemodialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- MK2578 1 mcg for every 600 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment every week (QW).
  Interventions: Drug: MK2578 1mcg for every 600 Units (U) of Epogen® (epoetin alfa) received per week at Baseline
- 1 mcg of MK2578 for every 600 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment QM.
  Interventions: Drug: MK2578 1mcg for every 600 Units (U) of Epogen® (epoetin alfa) received per week at Baseline
- MK2578 1 mcg for every 350 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment QW.
  Interventions: Drug: MK2578 1 mcg for every 350 U of Epogen (epoetin alfa) received per week at Baseline
- 1 mcg of MK2578 for every 350 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment QM.
  Interventions: Drug: MK2578 1 mcg for every 350 U of Epogen (epoetin alfa) received per week at Baseline
- MK2578 1 mcg for every 200 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment QW.
  Interventions: Drug: MK2578 1 mcg for every 200 U of Epogen (epoetin alfa) received per week at Baseline
- 1 mcg of MK2578 for every 200 U of Epogen at Baseline (Experimental): Participants were randomized to receive treatment QM.
  Interventions: Drug: MK2578 1 mcg for every 200 U of Epogen (epoetin alfa) received per week at Baseline

INTERVENTIONS:
Drug: MK2578 1mcg for every 600 Units (U) of Epogen® (epoetin alfa) received per week at Baseline — MK2578 was to be administered intravenously (IV). Participants in Cohort 1 were to receive 1 mcg of MK2578 for every 600 U of Epogen (epoetin alfa) received per week at Baseline. Participants were to be randomized to every week (QW) or once every 4 weeks (QM) dosing schedules within each cohort.
  Arms: 1 mcg of MK2578 for every 600 U of Epogen at Baseline; MK2578 1 mcg for every 600 U of Epogen at Baseline
Drug: MK2578 1 mcg for every 350 U of Epogen (epoetin alfa) received per week at Baseline — MK2578 was to be administered IV. Participants in Cohort 2 were to receive 1 mcg of MK2578 for every 350 U of Epogen (epoetin alfa) received per week at Baseline. Participants were to be randomized to QW or QM dosing schedules within each cohort.
  Arms: 1 mcg of MK2578 for every 350 U of Epogen at Baseline; MK2578 1 mcg for every 350 U of Epogen at Baseline
Drug: MK2578 1 mcg for every 200 U of Epogen (epoetin alfa) received per week at Baseline — MK2578 was to be administered IV. Participants in Cohort 3 were to receive 1 mcg of MK2578 for every 200 U of Epogen (epoetin alfa) received per week at Baseline. Participants were to be randomized to QW or QM dosing schedules within each cohort.
  Arms: 1 mcg of MK2578 for every 200 U of Epogen at Baseline; MK2578 1 mcg for every 200 U of Epogen at Baseline

SUMMARY:
This study will evaluate the efficacy and safety of intravenous MK2578, given as maintenance treatment for renal anemia in chronic kidney disease patients on dialysis who were previously receiving erythropoietin stimulating agents.

DETAILED DESCRIPTION:
This study consists of a 12-week base study (MK2578-003-AM03) and an optional 40-week extension study (MK2578-003-EXT12). Participants who complete 12 weeks of treatment in the base study will enter the extension on the most recent dose administered in the base study or a newly adjusted dose, if adjustment is required to bring Hg levels within range. Participants' doses of MK2578 will be adjusted upward or downward during the extension study to maintain Hb in the range of 10-12 g/dL.

ELIGIBILITY:
Inclusion Criteria:

Base Study:

* Patient is male or is a female who either cannot have children or who agrees to use appropriate contraceptive measures
* Patient has been on hemodialysis for at least 6 months when informed consent is signed
* Patient has received intravenous epoetin alfa or epoetin beta for a least 6 months when the informed consent is signed

Extension Study:

* Patient completed the base study through Week 12
* Patient tolerated MK2578 and demonstrated compliance with study procedures

Exclusion Criteria:

* Patient has a life expectancy of less than 6 months
* Patient is scheduled for a kidney transplant within the next 6 months
* Patient has had a blood transfusion within 12 weeks of screening
* Patient has had major surgery within 12 weeks of screening or plans to have surgery
* Patient has Human Immunodeficiency Virus (HIV)
* Patient has history of blood dyscrasia, hematologic disorders or any other disease known to cause anemia
* Patient has severe congestive heart failure (CHF)
* Patient has a history of malignant cancer, except certain skin or cervical cancers
* Patient has a history of grand mal seizures within the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 46 centers (9 centers in Bulgaria, 27 in United States, 3 in Romania, 4 in Italy, and 3 in Poland).
Pre-assignment Details: At randomization, participants received either MK2578 or matching placebo on Day 1 and crossed over to the alternate treatment at the next dialysis treatment on Day 3.
Groups:
- MK2578 1mcg/600 U or 1 mcg/350 U QW: MK2578 was administered intravenously (IV) QW. Participants were randomized to receive 1 mcg of MK2578 for every 350 Units (U) of Epogen (epoetin alfa) received per week at Baseline.
- MK2578 1mcg/600 U or 1 mg/350 U QM: MK2578 was administered IV QM. Participants were randomized to receive 1 mcg of MK2578 for every 600 Units (U) of Epogen (epoetin alfa) or 350 units of Epogen (epoetin alpha) received per week at Baseline.
Period: Overall Study
Arm/Group | MK2578 1mcg/600 U or 1 mcg/350 U QW | MK2578 1mcg/600 U or 1 mg/350 U QM
Started | 20 | 19
Completed | 8 | 9
Not Completed | 12 | 10
Not completed — Study terminated by sponsor | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- MK2578 1mcg/600U QW; MK2578 1mcg/350U QW: MK2578 IV administered QW.
- MK2578 1mcg/600U QM; MK2578 1mcg/350U QM: MK2578 IV administered QM.
- Total: Total of all reporting groups
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM | Total
Number analyzed (Participants) | 16 | 15 | 4 | 4 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (14.29) | 51.7 (10.22) | 58.0 (8.91) | 60.5 (4.51) | 51.0 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 3 | 3 | 24
  Male | 6 | 7 | 1 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hg) Level at Week 4
Time Frame: 4 weeks
Population: Full analysis set
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- MK2578 1mcg/600U QW: MK2578 IV was administered QW. Participants were randomized to receive 1 mcg of MK2578 for every 600 Units (U) of Epogen (epoetin alfa) received per week at Baseline.
- MK2578 1mcg/600U QM: MK2578 IV was administered QM. Participants were randomized to receive 1 mcg of MK2578 for every 600 U of Epogen (epoetin alpha) received per week at Baseline.
- MK2578 1mcg/350U QW: MK2578 IV was administered QW. Participants were randomized to receive 1 mcg of MK2578 for every 350 U of Epogen (epoetin alpha) received per week at Baseline.
- MK2578 1mcg/350U QM: MK2578 IV was administered QM. Participants were randomized to receive 1 mcg of MK2578 for every 350 U of Epogen (epoetin alpha) received per week at Baseline.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 16 | 14 | 1 | 1
g/dL | -0.6 (0.8) | -0.7 (1.0) | -1.0 (NA) — Only one patient was included in this analysis, thus the SD is not calculated. | -1.0 (NA) — Only one patient was included in this analysis, thus the SD is not calculated.

2. Primary Outcome: Number of Participants With Composite Events of Death, Myocardial Infarction (MI), and Cerebrovascular Accident (CVA)
Time Frame: 12 weeks
Measure: Number; unit: Participants
Groups:
- MK2578 1mcg/600U QW: MK2578 IV was administered QW. Participants were randomized to receive 1 mcg of MK2578 for every 600 U of Epogen (epoetin alpha) received per week at Baseline.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 16 | 15 | 4 | 4
Participants | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Composite Events of Transfusion-Related Adverse Experiences
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 16 | 15 | 4 | 4
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Composite Events of Infusion Reactions
Time Frame: 12 weeks
Measure: Number; unit: Participants
Groups:
- MK2578 1mcg/600 QM: MK2578 IV was administered QM. Participants were randomized to receive 1 mcg of MK2578 for every 600 U of Epogen (epoetin alpha) received per week at Baseline.
- MK2578 1mcg/350U QM: MK2578 IV was administered QM.Participants were randomized to receive 1 mcg of MK2578 for every 350 U of Epogen (epoetin alpha) received per week at Baseline.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600 QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 16 | 15 | 4 | 4
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Events of Death, MI, CVA, Peripheral Vascular Thromboses, Vascular Access Thrombosis, Congestive Heart Failure (CHF), Hypertension, Seizure, or Pure Red Cell Aplasia
Time Frame: 12 weeks
Measure: Number; unit: Participants
Groups:
- MK2578 1mcg/350U QW: MK2578 IV was administered QW. Participants were randomized to receive 1 mcg of MK2578 for every U of Epogen (epoetin alpha) received per week at Baseline.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 16 | 15 | 4 | 4
Participants
  Death | 0 | 0 | 0 | 0
  MI | 0 | 1 | 0 | 0
  CVA | 0 | 0 | 0 | 0
  Peripheral vascular thromboses | 0 | 0 | 0 | 0
  Vascular access thrombosis | 0 | 0 | 1 | 0
  CHF | 0 | 0 | 0 | 0
  Hypertension | 1 | 1 | 0 | 0
  Seizure | 0 | 0 | 0 | 0
  Pure red cell aplasia | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Confirmed, Treatment Emergent Antibodies to MK2578
Time Frame: 12 weeks
Population: Immunogenicity assays for antibodies to MK2578 were not performed due to early study termination.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK2578 1mcg/350U QM
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Hg Level at Week 12
Time Frame: 12 weeks
Population: Full analysis set; due to study termination participants in the MK2578 1mcg/350U QW and MK2578 1mcg/350U QM were not analyzed.
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- MK2578 1mcg/600U QW: MK3578 IV was administered QW. Participants were randomized to receive 1 mcg of MK-2578 for every 600 U of Epogen (epoetin alpha) received per week at Baseline.
- MK2578 1mcg/600U QM: MK2578 IV was administered QM. Participants were randomized to receive 1 mcg of MK2578 for every 600 Units (U) of Epogen (epoetin alfa) received per week at Baseline.
- MK2578 1mcg/350U QW: MK2578 IV was administered QW. Participants were randomized to receive 1 mcg of MK2578 for every 350 Units (U) of Epogen (epoetin alfa) received per week at Baseline.
- MK-2578 1mcg/350U QM: MK2578 IV was administered QM. Participatns were randomized to receive 1 mcg of MK2578 for every 350 Units (U) of Epogen (epoetin alpha) received per 4 weeks at Baseline.
Arm/Group | MK2578 1mcg/600U QW | MK2578 1mcg/600U QM | MK2578 1mcg/350U QW | MK-2578 1mcg/350U QM
Number analyzed (Participants) | 6 | 11 | 0 | 0
g/dL | -0.1 (1.4) | -0.5 (1.4) |  |

ADVERSE EVENTS:
Groups:
- MK2578 QW: MK2578 IV administered once weekly.
- MK2578 QM: MK2578 IV administered once every 4 weeks.
Arm/Group | MK2578 QW | MK2578 QM
Serious Adverse Events (participants affected / at risk) | 1/20 | 2/19
Other Adverse Events (participants affected / at risk) | 9/20 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK2578 QW (N=20) | MK2578 QM (N=19)
Acute mycoardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK2578 QW (N=20) | MK2578 QM (N=19)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal cyst (Endocrine disorders) | 0 (0) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Ultrasound pelvis abnormal (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Renal vein thrombosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Brachiocephalic vein stenosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Cohort 3 (MK2578 1mcg/200U) was not initiated because the study was prematurely

terminated by the sponsor. All randomized participants received at least one dose of study medication. Data presented are for Cohort 1 and Cohort 2, where applicable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.